CLINICAL TRIAL: NCT05345366
Title: The Impact of CITED2 on Collateral Circulation and Early Neurological Functional Outcome for Ischemic Stroke by Critically Regulating HIF-1α-VEGF Pathway
Brief Title: The Correlation Between CITED2 and Collateral Circulation in Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021LX0027-GC
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2022-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the good collateral group
  Interventions: Other: non-applicable
- the poor collateral group
  Interventions: Other: non-applicable

INTERVENTIONS:
Other: non-applicable — non-applicable

SUMMARY:
Evaluating the collateral circulation of acute ischemic stroke (AIS) mainly depends on the imaging examination. At present, there is no effective and sensitive biomarker for collateral circulation. Thus, the research objective was to evaluate the predicting role of the CBP/P300-interacting transactivator with Glu/Asp-rich C-terminal domain 2 Ratio (CITED2) from peripheral blood mononuclear cells in the collateral circulation of AIS. We classified the AIS patients into two groups (the good collateral group and the poor collateral group) by DWI-ASPECTS score. The western blot was applied to test the protein expression of vascular endothelial growth factor (VEGF) and CITED2. Then, we collected other clinical data. Binary logistic regression analysis between collateral circulation and clinical data was performed. Finally, Receiver operating characteristic (ROC) curve analysis was used to explore the predictive value of the CITED2.

ELIGIBILITY:
Inclusion Criteria:

* the first-time onset or previous stroke with mRS score ≤1, and the onset time less than 3 days without intravenous thrombolysis or endovascular therapy ;

  * age range of 18 to 80 years old;

    * patients with a clinical diagnosis of acute ischemic stroke; ④ NIHSS score ≥4; ⑤ patients volunteer to participate in this study and signed a written informed consent

Exclusion Criteria:

* ①the patients with AIS combined with other diseases that may affect the CITED2 and VEGF expression, such as acute myocardial infarction, peripheral artery occlusion disease and congenital heart defect;

  * the patients exhibited serious heart, live or kidney diseases; ③disturbance of consciousness or mental illness; ④ patients with tumor; ⑤ pregnant and lactating patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were diagnosed with acute ischemic stroke in the neurology department of our hospital from November 2020 to November 2023.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
CITED2 | within 24 hours after hospitalization
  western blot/ELISA
VEGF | within 24 hours after hospitalization
  western blot/ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lu M, Liu Y, Xian Z, Yu X, Chen J, Tan S, Zhang P, Guo Y. VEGF to CITED2 ratio predicts the collateral circulation of acute ischemic stroke. Front Neurol. 2022 Sep 30;13:1000992. doi: 10.3389/fneur.2022.1000992. eCollection 2022. PMID 36247751